CLINICAL TRIAL: NCT06022965
Title: Geriatric Assessment (GA)-Driven Interventions With Supportive Care (The GAIN-S Trial): Telemedicine to Increase Goal Concordant Care for Older Adults With Cancer in the Community
Brief Title: Telemedicine for Improvement of Care for Older Adults With Cancer in the Underserved Community, The GAIN-S Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22343; NCI-2023-05945 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22343 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-08-21; First posted 2023-09-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Geriatric Assessment; Palliative Care; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM I (GAIN-S) (Experimental): Patients complete the CARG-GA at baseline and 3 months and receive GA-based interventions using telemedicine over 6 months.
  Interventions: Other: Best Practice; Other: Comprehensive Geriatric Assessment; Other: Electronic Health Record Review; Other: Questionnaire Administration; Other: Supportive Care; Other: Telemedicine
- ARM II (SOC) (Active Comparator): Receive SOC over the first 3 months, then switch to receive GA-based interventions using telemedicine for the following 3 months.
  Patients complete the CARG-GA at baseline and 3 months and receive SOC over 6 months.
  Interventions: Other: Best Practice; Other: Comprehensive Geriatric Assessment; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive SOC
  Other Names: standard of care; standard therapy
Other: Comprehensive Geriatric Assessment — Complete CARG-GA
Other: Electronic Health Record Review — Ancillary studies
Other: Questionnaire Administration — Ancillary studies
Other: Supportive Care — Receive GA-based interventions
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: ARM I (GAIN-S)
Other: Telemedicine — Receive GA-based interventions via telemedicine
  Other Names: Telehealth
  Arms: ARM I (GAIN-S)

SUMMARY:
This clinical trial evaluates whether geriatric assessment-driven interventions with supportive care (GAIN-S) using telemedicine can be used to identify areas of vulnerability (weakness) in older adults with cancer and guide interventions to assist the patient and the healthcare team in the underserved community. The majority of patients diagnosed with cancer are over age 65 years, yet most cancer treatments are developed and tested in a younger population. Therefore, older patients with cancer are less likely to be offered standard treatments because of the concern regarding side effects. Geriatric assessment (GA) is a multi-dimensional health assessment tool combining patient reported and objective (unbiased) results. There is no standard tool that can identify which older adults will be more likely to have side effects from cancer treatment. Telemedicine is a way to provide healthcare services (including consultations, education, care management and treatment) in which the health care provider is at a distant site. The goal of this project is to use telemedicine to identify areas of vulnerability/weakness in older adults with cancer using a patient assessment, and to identify the potential referrals to a multi-specialty team based on patient assessment results. Information gathered from this study may help researchers learn whether GAIN-S can be performed using telemedicine and lead to improvement in care for older adults compared to standard of care (SOC) in the underserved community.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To implement Geriatric Assessment-driven interventions with supportive care (GAIN-S) through telemedicine to:

Ia. To improve communication between the primary care team (oncologist, nurses) and patients and caregivers in a remote community setting to increase prognostic discussions and goal concordant care; Ib. To improve cost-saving in older patients with cancer.

SECONDARY OBJECTIVES:

I. Determine whether GAIN-S implemented in a community setting will lead to a decrease in treatment toxicity.

II. To examine whether GAIN-S intervention will lead to improvement in hospitalizations, dose delays, dose reduction and discontinuation.

III. To compare patient satisfaction using the "Was It Worth It" (WIWI) between the 2 arms at the 3 and/or 6-month timepoint.

IV. To compare patient preferences at baseline, using the validated patient-defined treatment preference and goals measures between the 2 arms and longitudinal change, at 3 and/or 6-month timepoint.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (GAIN-S): Patients complete the Cancer and Aging Research Group-Geriatric Assessment (CARG-GA) at baseline and 3 months and receive GA-based interventions using telemedicine over 6 months.

ARM II (SOC): Patients complete the CARG-GA at baseline and 3 months and receive SOC over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant.
* Patient's physician must agree for patient participation.
* Ability to read English, Spanish, or Chinese. Other languages will be acceptable with site principal investigator (PI) agreement if surveys are available, and language does not preclude completing study procedures.
* Age: >=65 years at the time of enrollment.
* Diagnosis of stage I-IV cancer.
* Scheduled to start a new therapy (chemotherapy, immunotherapy, or targeted therapy).

Exclusion Criteria:

* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2027-01-24 (Estimated); Study Completion 2027-01-24 (Estimated)

PRIMARY OUTCOMES:
Rate of advance directive (AD) completion | At start of treatment and 3 months after treatment initiation
  Will be assessed using medical chart review. Chi-square test will be used to compare the proportions of AD completion between the two arms.
Number of documented conversations. | At start of treatment and 3 months after treatment initiation
  Will be assessed using medical chart review. T-test will be used to compare the mean number of documented conversations between the two arms.
Direct inpatient cost | At 3 and 6-months after treatment initiation
  Will log transformed and Z-score test will be used to compare the mean costs of the two arms. Chi-square test will be used to compare number of patients with short verse (vs.) long stay and Intensive Care Unit (ICU) admission between the two arms.

SECONDARY OUTCOMES:
Decrease in treatment toxicity | At 3 months after randomization
  Will be described using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and will examine toxicities by grade and type. Chi-square test will be used to compare proportion of patients with grade 3-5 toxicity, dose modifications including dose change, dose delay, discontinuation as well as hospitalization, consider treatment worthwhile between two arms.
Proportion of patients with dose modifications | Up to 6 months
  Defined as delays and dose change experienced by patients for each cohort at each cycle. The reason for dose modifications will be noted and attributed as possibly, probably, or definitely related to treatment. Chi-square test will be used to compare proportion of patients with grade 3-5 toxicity, dose modifications including dose change, dose delay, discontinuation as well as hospitalization, consider treatment worthwhile between two arms.
Patient satisfaction using the "Was It Worth It" (WIWI) | At 3 and/or 6-months after treatment initiation
  Patient satisfaction assessed as whether patients found treatment worthwhile using the "Was it Worth it" (WIWI) questionnaire.
  T-test will be used to compare satisfaction rating between the two arms. Chi-square test will be used to compare proportion of patients consider treatment worthwhile between the two groups.
Patient preferences and goals | At baseline, 3 and/or 6 months after treatment initiation
  Patient-Defined Treatment Preferences and Goals will be measured utilizing the Health Outcomes Questionnaire, Now vs Later Tool and Attitude Scale. Will use the validated patient-defined treatment preference and goals measures between the 2 arms and longitudinal change. Descriptive statistics and plots will be used to describe and compare of longitudinal changes in patient preferences and goals will be plotted.
Association of Community Cancer Centers (ACCC) Geriatric Oncology Gap Assessment Tool | Baseline and at the end of study (36 months)
  The tool's name is: Association of Community Cancer Centers: Geriatric Oncology Gap Assessment Tool Scoring for the tool is based on a 1-4 scale with Level 4 representing the optimal practice.
  Prior to study initiation, each site will be quantitatively evaluated utilizing the evidence-based ACCC Geriatric Oncology Gap Assessment tool; each site would be reassessed at the end of the study. This tool will provide an evidence-based assessment to evaluate the current geriatric oncology efforts at each site and guide future steps for improvement to these services.

CONTACTS AND LOCATIONS:
Overall Officials: William Dale, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope Upland, Upland, California